CLINICAL TRIAL: NCT07355049
Title: The Effect of Intravenous Dexmedetomidine Versus Intravenous Lidocaine on the Emergence Agitation After Endoscopic Sinus Surgery. A Prospective, Randomized, Double-blind Controlled Trial.
Brief Title: The Effect of Dexmedetomidine Versus Lidocaine on Emergence Agitation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Khaled Eid Tolba Abo Elwa, Doctor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: M786
Record Dates: First submitted 2025-11-15; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Emergence Agitation
Keywords: Emergence agitation; Intravenous dexmedetomidine; Endoscopic sinus surgery; Intravenous lidocaine
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Active Comparator): Active comparator group Group (L) recieves IV lidocaine 1.5mg/kg slowly before induction of anesthesia then lidocaine infusion starts at a rate of 2mg/kg/h
  Interventions: Drug: Lidocaine
- Group D (Active Comparator): Active comparator group (D) recieves IV dexmedetomidine bolus dose of 1mcg/kg over 10 minutes before induction of anesthesia followed by continous infusion at 0.4mcg/kg/h until the end of surgery
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Group (D) recieves Dexmedetomidine bolus 1mcg/kg over 10 minutes before induction of anesthesia followed by continous infusion at 0.4 mcg/kg/h until the end of surgery
  Arms: Group D
Drug: Lidocaine — Group (L) recieves IV lidocaine 1.5 mg/kg slowly before induction of anesthesia then lidocaine infusion starts at a rate of 2mg/kg/h
  Arms: Group L

SUMMARY:
The effect of intravenous dexmedetomidine versus intravenous lidocaine on the emergence agitation after endoscopic sinus surgery.

DETAILED DESCRIPTION:
Endoscopic sinus surgery (ESS) is a common operation for patients with chronic rhinosinusitis with nasal polyps (CRSwNP) when medical therapy alone is insufficient .

Early recovery from general anesthesia is accompanied by agitation, confusion, disorientation, and violent behavior, which is known as Emergence Agitation (EA). This post-anesthetic issue occurs in the early stages of General Anesthesia (GA) recovery, posing challenges in terms of both patient recovery delay and the complexities associated with assessment and management.

The incidence of EA varies, from approximately 0.25% to 90.5%, with age, assessment tool used, definitions, anesthetic techniques, type of surgery, and time of EA assessment during recovery .

Because the airway is contaminated with blood and the nasal airway is closed with surgical packs. ENT surgery is linked to a higher incidence of emerging agitation after nasal surgery.

Although EA is commonly self-limited and happens within the first 30 min of stay in a postanesthesia care unit (PACU) and also can lead to disconnection of monitoring devices or intravenous catheters, physical damage, falling, increase in the risk of bleeding, and self-extubation .

Several pharmacological methods have been used to mitigate EA, including opioid (fentanyl, remifentanil), propofol, benzodiazepine (midazolam), α2- aderenoreceptor agonist (clonidine, dexmedetomidine), and N-methy-d-aspar- tate (NMDA) receptor antagonist (ketamine, magnesium sulfate) administration.

Lidocaine is an amino amide-type short-acting local anesthetic (LA). It has a short half-life, and a favorable safety profile, and is therefore the LA of choice for continuous IV administration. Systemic lidocaine has been shown to be an effective adjunct strategy to reduce postoperative pain.

Dexmedetomidine is known as a highly selective α (2)-adrenoceptor agonist with sedative, anxiolytic, sympatholytic, and analgesic-sparing effects, which causes minimal depression of the respiratory function.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-60
* ASA Physical Status I or II
* Elective endoscopic sinus surgery under general anesthesia .

Exclusion Criteria:

* Refusal to participate
* Mental retardation or inability to communicate
* Allergy to anesthetics or study medications .
* Chronic use of beta blockers .
* significant hepatic, neurologic, cardiovascular or respiratory disease .
* BMI>35 kg/m2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-21 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence agitation (EA) . | Immediate after extubation
  Incidence of emergence agitation (EA) as measured by Richmond Agitation Sedation Scale (RASS) .

SECONDARY OUTCOMES:
heart rate (beats per minute ) | baseline ( preoperative )
  heart rate (beats per minute ) was measured using standard ECG monitoring
heart rate (beats per minute ) | after 30 minutes ( intraoperative)
  heart rate (beats per minute ) was measured using standard ECG monitoring
heart rate (beats per minute) | after 60 minutes ( intraoperative )
  heart rate (beats per minute ) was measured using standard ECG monitoring
heart rate (beats per minute) | 0 hour postoperative
  heart rate (beats per minute ) was measured using standard ECG monitoring
heart rate (beats per minute) | 1 hour postoperative
  heart rate (beats per minute ) was measured using standard ECG monitoring
heart rate (beats per minute) | 3 hours postoperative
  heart rate (beats per minute ) was measured using standard ECG monitoring
heart rate (beats per minute) | 6 hours postoperative
  heart rate (beats per minute ) was measured using standard ECG monitoring
heart rate (beats per minute) | 12 hours postoperative
  heart rate (beats per minute ) was measured using standard ECG monitoring
heart rate (beats per minute) | 24 hours postoperative
  heart rate (beats per minute ) was measured using standard ECG monitoring
Mean arterial blood pressure (mmHg) | baseline ( preoperative )
  MAP ( mmHg) was measured using standard non-invasive blood pressure monitoring .
Mean arterial blood pressure (mmHg) | after 30 minutes ( intraoperative )
  MAP ( mmHg) was measured using standard non-invasive blood pressure monitoring .
Mean arterial blood pressure (mmHg) | after 60 minutes ( intraoperative )
  MAP ( mmHg) was measured using standard non-invasive blood pressure monitoring .
Mean arterial blood pressure (mmHg) | 0 hour post operative
  MAP ( mmHg) was measured using standard non-invasive blood pressure monitoring .
Mean arterial blood pressure (mmHg) | 1 hour post operative
  MAP ( mmHg) was measured using standard non-invasive blood pressure monitoring .
Mean arterial blood pressure (mmHg) | 3 hour post operative
  MAP ( mmHg) was measured using standard non-invasive blood pressure monitoring .
Mean arterial blood pressure (mmHg) | 6 hour post operative
  MAP ( mmHg) was measured using standard non-invasive blood pressure monitoring .
Mean arterial blood pressure (mmHg) | 12 hour post operative
  MAP ( mmHg) was measured using standard non-invasive blood pressure monitoring .
Mean arterial blood pressure (mmHg) | 24 hour post operative
  MAP ( mmHg) was measured using standard non-invasive blood pressure monitoring .
Peripheral oxygen saturation (SpO2, %) | baseline ( preoperative )
  Peripheral oxygen saturation (SpO2, %) was measured using pulse oximetry
Peripheral oxygen saturation (SpO2, %) | after 30 minutes ( intraoperative )
  Peripheral oxygen saturation (SpO2, %) was measured using pulse oximetry
Peripheral oxygen saturation (SpO2, %) | after 60 minutes ( intraoperative)
  Peripheral oxygen saturation (SpO2, %) was measured using pulse oximetry
Peripheral oxygen saturation (SpO2, %) | 0 hour post operative
  Peripheral oxygen saturation (SpO2, %) was measured using pulse oximetry
Peripheral oxygen saturation (SpO2, %) | 1 hour post operative
  Peripheral oxygen saturation (SpO2, %) was measured using pulse oximetry
Peripheral oxygen saturation (SpO2, %) | 3 hour post operative
  Peripheral oxygen saturation (SpO2, %) was measured using pulse oximetry
Peripheral oxygen saturation (SpO2, %) | 6 hour post operative
  Peripheral oxygen saturation (SpO2, %) was measured using pulse oximetry
Peripheral oxygen saturation (SpO2, %) | 12 hour post operative
  Peripheral oxygen saturation (SpO2, %) was measured using pulse oximetry
Peripheral oxygen saturation (SpO2, %) | 24 hour post operative
  Peripheral oxygen saturation (SpO2, %) was measured using pulse oximetry
Postoperative pain score | 0, 1 h(hour), 3h, 6h, 12h, 24h postoperatively
  Postoperative pain was assessed using the Numeric rating scale (NRS) , ranging from 0 ( no pain ) to 10 ( worst imaginable pain )
Incidence of adverse events | first 24 hours postoperative
  Incidence of adverse events including postoperative nausea&vomiting , allergy , bradycardia (HR<50) , hypotension (MAP decreases by >20%) , desaturation ( SpO2<92%)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled E Tolba, MBBCH, Principal Investigator
Locations (1):
- FayoumU, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mohkamkar M Bs, Farhoudi F Md, Alam-Sahebpour A Md, Mousavi SA Md, Khani S PhD, Shahmohammadi S BSc. Postanesthetic Emergence Agitation in Pediatric Patients under General Anesthesia. Iran J Pediatr. 2014 Apr;24(2):184-90. PMID 25535538
- [Result] Lourijsen ES, Reitsma S, Vleming M, Hannink G, Adriaensen GFJPM, Cornet ME, Hoven DR, Videler WJM, Bretschneider JH, Reinartz SM, Rovers MM, Fokkens WJ. Endoscopic sinus surgery with medical therapy versus medical therapy for chronic rhinosinusitis with nasal polyps: a multicentre, randomised, controlled trial. Lancet Respir Med. 2022 Apr;10(4):337-346. doi: 10.1016/S2213-2600(21)00457-4. Epub 2022 Jan 7. PMID 35012708